CLINICAL TRIAL: NCT02477462
Title: Identification of Inflammatory and Fibrotic Biomarkers in PBC and NAFLD Patients
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 703097
Record Dates: First submitted 2015-06-10; First posted 2015-06-22 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ambulatory Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Biospecimens will include serum, plasma, DNA, and RNA. In 20 subjects liver biopsies will be performed and retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Primary Biliary Cirrhosis: Subjects meeting internationally accepted criteria for the diagnosis of primary biliary cirrhosis
  Interventions: Other: Clinic visit
- Control: Subjects without evidence of primary biliary cirrhosis, liver disease, or inflammatory condition who are of similar age and sex distribution to the Primary Biliary Cirrhosis group
  Interventions: Other: Baseline visit

INTERVENTIONS:
Other: Clinic visit — Blood draw every 3 months; quality of life surveys and imaging annually
  Groups: Primary Biliary Cirrhosis
Other: Baseline visit — Blood draw and quality of life surveys
  Groups: Control

SUMMARY:
Primary biliary cirrhosis (PBC) is a progressive autoimmune disease of biliary epithelial cells resulting in biliary cirrhosis. PBC is characterized by a 90% female predominance, high titers of serum anti-mitochondrial autoantibodies (AMA) directed against the pyruvate dehydrogenase complex E2 subunit and evidence from both human and murine models suggests that T-cells, particularly cluster of differentiation (CD) 8+ T cells, are key to the destruction of bile ducts. However, clinical trials of classic immunosuppressive drugs including corticosteroids, azathioprine, methotrexate, and tacrolimus have been largely unsuccessful in altering the disease course. This is a single center, prospective, non-treatment study of the role of immune responses in PBC patients.

Non-alcoholic fatty liver disease (NAFLD) and its more severe form, non-alcoholic steatohepatitis (NASH) are common, often "silent" liver diseases. NASH resembles alcoholic liver disease, but occurs in people who drink little or no alcohol. The major feature in NASH is fat in the liver, along with inflammation and fibrosis. NASH can be severe and can lead to cirrhosis and hepatocellular carcinoma. Ten to 20 percent of American have NAFLD with NASH affecting 2 to 5 percent of Americans.

DETAILED DESCRIPTION:
In this study, the investigators will prospectively collect demographic, clinical, and laboratory data and blood samples for research purposes on 45 PBC patients and 50 male and female NAFLD patients. PBC and NAFLD diagnosis and clinical status will be evaluated by magnetic resonance (MR) elastography, transient elastography (FibroScan®) and blood lab analysis including anti-mitochondrial antibodies (AMA), anti-nuclear antibodies (ANA), immunoglobulins, complete blood count (CBC), comprehensive metabolic panel (CMP) and coagulation measures). Additionally serum and blood will be obtained from the patients on the first visit and at months 3, 6, 9, 12, 15, 18, 21 & 24. Serum and blood samples will be used to measure serum cytokine abundance and transcriptome analysis. For comparison, 95 age (+/- 5 years) and sex-matched controls without PBC will be recruited for a clinical laboratory, cytokine, gene expression analysis. Control subjects will have blood drawn at a single time point.

ELIGIBILITY:
Inclusion Criteria for Primary Biliary Cirrhosis Group:

* PBC diagnosis based upon at least 2 of 3 criteria: AMA titer > 1:40; Alkaline phosphatase > 1.5 times the upper limit of normal (ULN) for at least 6 months; and Liver biopsy findings consistent with PBC
* 18 years of age and older.

Exclusion Criteria:

* Presence of other concomitant liver diseases including viral hepatitis, primary sclerosing cholangitis (PSC), alcoholic liver disease, Wilson's disease, hemochromatosis, or Gilbert's syndrome.
* Prior liver transplantation
* Use of immunosuppressants within 6 months of Day 0, including azathioprine, prednisone, prednisolone, budesonide, cyclosporine, tacrolimus, methotrexate, or mycophenolate mofetil.
* Use of biologic agents including anti-cell and anti-cytokine therapies within 12 months.

Inclusion Criteria for Control Subjects

* Absence of liver disease or inflammatory conditions
* 18 years of age and older.

Exclusion Criteria for Control Subjects

* Presence of concomitant liver diseases including PBC, viral hepatitis, PSC, alcoholic liver disease, Wilson's disease, hemochromatosis, or Gilbert's syndrome.
* Prior liver transplantation
* Use of immunosuppressants within 6 months, including azathioprine, prednisone, prednisolone, budesonide, cyclosporine, tacrolimus, methotrexate, or mycophenolate mofetil.
* Use of biologic agents including anti-cell and anti-cytokine therapies within 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Confirmed PBC diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-05; Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Phenotypic Analysis | 2 years
  Comparison of PBC phenotypes defined by alkaline phosphatase response to treatment and degree of fibrosis determined by transient elastography. In addition, Principle component analysis (PCA) and non-negative matrix factorization (NMF) will be used to identify phenotypic subject stratification utilizing both cytokine and gene expression data at baseline. The alkaline phosphatase (ALP) will be compared between these classes to determine if there is an association between classes.

SECONDARY OUTCOMES:
Liver Imaging Analysis | 2 years
  Transient elastography (FibroScan) and MR elastography will provide a measurement of liver stiffness. The liver stiffness metrics will be tabulated for each of the three time points and assessed for change.
Phlebotomy Injuries | 2 years
  Number of injuries occurring as a result of phlebotomy during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Bowlus, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States